CLINICAL TRIAL: NCT02325960
Title: A Comparison of Exenatide and Insulin Glargine on Glycemic Variability in T2DM Patients Inadequately Controlled With Metformin Monotherapy
Brief Title: A Comparison of Exenatide and Insulin Glargine
Status: Completed | Phase: Phase 4 | Type: Interventional
Sponsor: The Affiliated Nanjing Drum Tower Hospital of Nanjing University Medical School (Other)
Responsible Party: Principal Investigator, Dalong Zhu, Chief physician, The Affiliated Nanjing Drum Tower Hospital of Nanjing University Medical School
Allocation: Randomized | Model: Parallel | Masking: None | Purpose: Treatment
Other Study IDs: ISSEXEN0034
Record Dates: First submitted 2014-10-29; First posted 2014-12-25 (Estimated); Last update posted 2017-02-23 (Actual); Status verified 2017-02

CONDITIONS: Type 2 Diabetes
Keywords: exenatide; insulin glargine
MeSH Terms: conditions — Diabetes Mellitus, Type 2 | interventions — Exenatide; Insulin Glargine

STUDY DESIGN:
Oversight: Data Monitoring Committee: Yes

ARMS (2):
- exenatide (Active Comparator): 5 μg BID for the first 4 weeks of treatment and 10 μg thereafter
  Interventions: Drug: exenatide; Drug: Insulin glargine
- Insulin glargine (Active Comparator): ≥8 IU QD, and titrate based on a dosing algorithm targeting FPG <6.1 mmol/L. Titration is only allowed in first 4 weeks.
  Interventions: Drug: exenatide; Drug: Insulin glargine

INTERVENTIONS:
Drug: exenatide — 5 μg BID for the first 4 weeks of treatment and 10 μg thereafter.
  Other Names: Byetta.Lilly
Drug: Insulin glargine — ≥8 IU QD, and titrate based on a dosing algorithm targeting FPG <6.1 mmol/L. Titration is only allowed in first 4 weeks.
  Other Names: Lantus,Sanofi Aventis

SUMMARY:
This is a 16-week, Single-center, Randomized, Open Label, Parallel Controlled Group Comparison of the Comprehensive Glycemic Control of Exenatide and Insulin Glargine on Type 2 Diabetes Patients Inadequately Controlled With Metformin Monotherapy.

DETAILED DESCRIPTION:
Screening will be made to select eligible patients, then 44 patients receiving a stable dose of metformin (≥1500 mg daily) will be randomized (1:1) to receive exenatide or insulin glargine for 16 weeks. Exenatide will be administered twice daily by subcutaneous injection 30- 60 minutes before breakfast and dinner; the dose was 5 μg twice-daily for the first 4 weeks of treatment and 10 μg thereafter. Insulin glargine will be administered once daily at bedtime by subcutaneous injection. The dose of insulin glargine will initiate at ≥8 IU once-daily, and titrate based on a dosing algorithm targeting fasting blood glucose (FPG)<6.1 mmol/L. Titration is only allowed in first 4 weeks. At the end of the study, data will be collected and analyzed.

ELIGIBILITY:
Inclusion Criteria:

1. Provision of informed consent prior to any study specific procedures
2. Type2 diabetic patients had been on stable, maximum tolerated doses of metformin (≧1500mg/d, ≧8 weeks)
3. Male or female age ≧ 18 years and ≦70 years old
4. HbA1c ≧7.0 and ≦10%
5. BMI ≧ 24 kg/m2

Exclusion Criteria:

1. Known or suspected allergy to trial products or related products.
2. Impaired renal function defined as serum-creatinine ≥ 1.5 mg/dl (≥ 133 umol/l).
3. Acute or chronic disease which may cause tissue hypoxia such as respiratory failure or shock.
4. Abnormal liver function, alanine transaminase or aspartate aminotransferase ≥ 3 fold normal upper limit, Total bilirubin ≥ 2 normal upper limit, acute alcohol intoxication, alcoholism.
5. Subjects has a clinically significant, active (or over the past 12 months) cardiovascular history (including a history of myocardial infarction (MI), arrhythmias or conduction delays on ECG, unstable angina, or decompensated heart failure (New York Heart Association-class Ⅲ and Ⅳ).
6. Proliferative retinopathy or muscular oedema requiring acute treatment.
7. Pregnant or positive pregnancy test at screening, nursing mother, or unwillingness to use adequate contraception (adequate contraceptive measures are sterilization, intrauterine device, oral contraceptives or barrier methods).
8. Treatment with systemic corticosteroids within the past two months prior to screening.
9. Type 1 diabetes mellitus.
10. Receipt of any investigational drug within 1 month prior to this trial.

Ages: 18 Years to 70 Years | Sex: All | Healthy Volunteers: No
Age Groups: Adult, Older Adult
Enrollment: 44 (Actual)
Dates: Start 2015-01; Primary Completion 2016-07 (Actual); Study Completion 2016-10 (Actual)

PRIMARY OUTCOMES:
Mean amplitude of glycemic excursions (MAGE) change from baseline by continuous glucose monitoring system (CGMS) | 1±3day；112±3d

SECONDARY OUTCOMES:
Glycemic variability | 1±3day；112±3d
  continuous overlapping net glycemic action (CONGA) and mean of daily differences (MODD)
Glucose control | -7±3d；112±3d；
  Glycosylated hemoglobin A 1c (HbA1c), FBG, postprandial blood glucose (PBG)
oxidative stress markers | 1±3d；28±3d；56±3d；84±3d；112±3d
  plasma concentrations of superoxide dismutase (SOD), malondialdehyde, 8-iso-prostaglandin-F2α (8-iso-PGF2α) and urine concentrations of 8-iso-PGF2α;
inflammatory markers | 1±3d；28±3d；56±3d；84±3d；112±3d
  plasma concentrations of interleukin-1(IL-1), interleukin-18(IL-18), adiponectin, toll-like receptor 4(TLR-4) and phosphorylated-nuclear factor-kappaB 65 (pNF-κB 65) in white blood cells
endothelial function | 1±3d；28±3d；56±3d；84±3d；112±3d
  plasma total nitric oxide synthase (tNOS), inducible nitric oxide synthase (iNOS), nitric oxide (NO)
beta-cell function and insulin resistance | 1±3d；112±3d；
  homeostasis model assessment-β, homeostasis model assessment -insulin resistance, plasma glucagon, body mass index (BMI), waist-hip ratio
body composition | 1±3d；112±3d
  fat mass, lean tissue, body weight, waist circumference

OTHER OUTCOMES:
Number of Participants with exenatide or insulin glargine adverse events as a measure of safety and tolerability: | -7±3d；1±3d；7±2d；14±3d；21±2d；28±3d；35±3d；56±3d；84±3d；112±3d
  hypoglycemia reaction; blood glucose lower than 3.1mmol/L; nausea, vomiting, diarrhea, anorexia or abdominal pain after exenatide subcutaneous injection.
Exploratory Objective assessed by the relationships between oxidative stress and inflammatory markers and MAGE | 1±3d；112±3d
  Whether there is linear correlation between oxidative stress markers and MAGE, and between inflammatory markers and MAGE, and correlation coefficient of each correlation

CONTACTS AND LOCATIONS:
Overall Officials: Dalong Zhu, MD PhD, Principal Investigator — the Affiliated Drum Tower Hospital of Nanjing University
Locations (1):
- at Division of Endocrinology, the Affiliated Drum Tower Hospital of Nanjing University, Nanjing, Jiangsu, China

IPD SHARING:
Plan to Share IPD: Undecided

REFERENCES:
- [Derived] Yin TT, Bi Y, Li P, Shen SM, Wang WM, Jiang C, Gao CX, Wang Y, Gao LJ, Zhu DL, Feng WH. Effects of exenatide versus insulin glargine on body composition in overweight and obese T2DM patients: a randomized controlled trial. Nutr Metab (Lond). 2018 Oct 1;15:67. doi: 10.1186/s12986-018-0295-6. eCollection 2018. PMID 30302121